CLINICAL TRIAL: NCT02585232
Title: Optimizing Dementia Care Through Collaborative Recovery Interventions
Brief Title: Optimizing Dementia Care
Acronym: ODeC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D1824-W
Record Dates: First submitted 2015-10-14; First posted 2015-10-23 (Estimated); Results first posted 2021-09-13 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Alzheimer's Disease; Dementia; Dementia, Vascular; Caregivers; Veterans
Keywords: Behavioral sciences; Counseling; Intervention Studies; Cognitive Behavioral Therapy; Telemedicine; Mindfulness
MeSH Terms: conditions — Alzheimer Disease; Dementia; Dementia, Vascular | interventions — Counseling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Care Consultation (CC) (Active Comparator): Care Consultation (CC): is an established telephone-based, empowerment intervention that uses coaching and emotional support to mobilize family caregivers and individuals with dementia through psychoeducation, resource referral, psychosocial support, and encouragement of informal and formal service use utilization. A computerized clinical tool called the Care Consultation Information System (CCIS) guides the care consultant through a standardized delivery of protocol components. Rather than a strong focus on assessment, this intervention is designed to quickly identify areas of unmet need through brief trigger questions called the "initial assessment" - much like an interview guide - which then immediately shapes development of concrete action plans.
  Interventions: Behavioral: Care Consultation (CC)
- Care Consultation + Counseling (CC+C) (Experimental): Care Consultation + Counseling (CC+C): is consistent with the original CC protocol in that the therapist partners with each dyad in a patient-centered way to prioritize unmet needs as identified during the CC initial assessment. Once this phase has been completed, typically within the first 2 sessions, the CC+C therapist will determine when to initiate counseling sessions targeting 8-10 domains of potential distress (grief, hostility, sexual intimacy, etc.). The counseling component of the CC+C intervention incorporates elements of existing manualized interventions that have been tailored for this population and follow a cognitive behavioral therapy framework.
  Interventions: Behavioral: Counseling (C); Behavioral: Care Consultation (CC)

INTERVENTIONS:
Behavioral: Counseling (C) — The counseling component incorporates elements of existing manualized interventions that have been tailored for this population and follow a cognitive behavioral therapy framework. Counseling sessions will be completed for 8-10 domains of potential distress (grief, hostility, sexual intimacy, etc.).
  Arms: Care Consultation + Counseling (CC+C)
Behavioral: Care Consultation (CC) — Care Consultation (CC): is an established telephone-based, empowerment intervention that uses coaching and emotional support to mobilize family caregivers and individuals with dementia through psychoeducation, resource referral, psychosocial support, and encouragement of informal and formal service use utilization. A computerized clinical tool called the Care Consultation Information System (CCIS) guides the care consultant through a standardized delivery of protocol components. Rather than a strong focus on assessment, this intervention is designed to quickly identify areas of unmet need through brief trigger questions called the "initial assessment," which then immediately shapes development of concrete action plans.

SUMMARY:
The purpose of this randomized controlled pilot study is to examine the preliminary effectiveness, feasibility, and potential treatment moderators (i.e., behavioral symptoms and spousal relationship status) of a newly developed intervention for individuals with dementia and their family caregivers that combines elements of the established care consultation (CC) approach with additional counseling modules (CC+C). Outcomes for Veterans with dementia and their family caregivers (e.g., depressive symptoms, care-related burden, quality of life, pleasant events, etc.) will be assessed after 6 months of treatment and again at 12 months.

DETAILED DESCRIPTION:
Background: Dementia affects over 7% of Veterans age 65 and above seeking care through the Veteran's Health Administration (VHA), amounting to one out of every eleven Veterans in some VISNs. The unique functional and behavioral impairments associated with Alzheimer's or a related dementia (ADRD) contribute substantially to psychological and physical morbidity of family caregivers and high rates of nursing home placement, with 60% of ADRD caregivers rating the emotional stress of caregiving as "high or very high," and over one third reporting depressive symptoms. Although numerous evidence-based interventions have been developed to reduce caregiver burden and improve mental health and functional outcomes of the person with dementia, a recent systematic review noted almost none of these interventions "make it off of the shelf" to be readily available in clinical settings. Care Consultation (CC) has emerged as a rare exception. CC is an evidence-based telephone intervention delivering psychoeducation, care coordination, and resource referrals in diverse areas such as safety and mental and behavioral health support. Yet CC's focus on coaching and support is inadequate for dyads experiencing high levels of distress. A stepped-intervention approach would address the VA's efficiency needs while allowing the flexibility for more resource-intensive additional counseling beyond the established CC framework when warranted by high dyad distress. This CDA-2 proposal would move such a dyadic intervention forward.

Objectives: 1) Manualize the integration of care consultation and counseling components (i.e., the CC+C intervention). CC+C is guided by a rehabilitation recovery-based conceptual model to address the most common high distress targets (e.g., relationship distress, Veteran or caregiver depression, anxiety, or pain) using patient-centered approaches. 2) Evaluate preliminary effectiveness and feasibility of the CC+C Intervention in a randomized controlled pilot study of distressed dyads to compare: a) the established CC intervention, to b) the CC+C intervention on Veteran and caregiver outcomes. 3) Conduct exploratory analyses of the CC+C intervention on Veteran long-term care placement at six and 12 months and examine two key treatment moderators (behavioral symptoms and spousal relationship status) that may impact intervention engagement and response to treatment.

The investigators hypothesize that: 1) Caregivers assigned to CC+C will have greater reductions in caregiver burden at 6 months than those assigned to CC alone. 2) Indicators of relationship strain (i.e., marital distress and/or mutuality) will show greater improvement in CC+C than CC at 6 months. 3) Gains in shared pleasant events, social engagement, and quality of life will be greater in CC+C than in CC alone at 6 months. 4) Participants with dementia in both groups will have reduced depressive symptoms at 6 months. The investigators will also explore the impact of the two interventions on rates of placement in long-term care facilities (such as nursing homes, VA Community Living Centers or other supportive living environments) at 6 and 12 months.

Methods: Ten modules combining successful elements from existing manualized therapies and exercises developed by the investigative team during the CDA1 period will be integrated with CC into a draft CC+C intervention manual. The manual will be finalized with input from the mentoring team and an Expert Advisory Panel for completeness, feasibility, and safety and risk considerations. Next 68 distressed Veterans with dementia and their family caregivers will be recruited and randomized to either the CC+C intervention group or the CC comparison group. Patient, caregiver, and relationship outcomes (e.g., burden, depressive symptoms, anxiety, quality of life, relationship distress) will be measured at baseline, 6 months, and 12 months. Treatment implementation and feasibility data will be collected.

Anticipated Impacts: The goal of this career development study is to acquire the knowledge, skills and experience necessary to successfully compete for an RR&D Merit Review Award evaluating a randomized controlled trial powered to establish efficacy and test effectiveness of the CC+C intervention. Rehabilitation-focused interventions that maximize functioning are essential for successful non-institutional VA dementia care in the future. Work completed during the CDA2 period will serve as a foundation for a career committed to this goal. The impact of this work will be realized when an efficacious and highly-accessible intervention, such as the telephone-based dyadic intervention being piloted, becomes available for aging Veterans and their families.

ELIGIBILITY:
Inclusion Criteria:

Veterans:

* Must be age 19 or older
* Must have a diagnosis of dementia or a related disorder
* Must live in the community (i.e. not in a VA Community Living Center, nursing home, or other facility)
* Must cohabitate with a caregiver
* Must have reliable access to a telephone
* Must be willing to consent to participate or provide assent in conjunction with proxy consent if their decision-making capacity is compromised

Caregivers:

* Must be age 19 or older
* Must self-identify as assisting with care for at least 8 hours/week
* Must be willing to consent to participate

Exclusion Criteria:

Veterans:

* Currently incarcerated
* Currently pregnant
* Dyads experiencing low levels of distress

Caregivers:

* Currently incarcerated
* Currently pregnant
* Experiencing severe cognitive impairment that would impair their ability to communicate during an interview
* Dyads experiencing low levels of distress

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2020-08-05 (Actual); Study Completion 2020-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle M Hilgeman, PhD, Principal Investigator — Tuscaloosa VA Medical Center, Tuscaloosa, AL
Locations (1):
- Tuscaloosa VA Medical Center, Tuscaloosa, AL, Tuscaloosa, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Judge KS, Bass DM, Snow AL, Wilson NL, Morgan R, Looman WJ, McCarthy C, Kunik ME. Partners in dementia care: a care coordination intervention for individuals with dementia and their family caregivers. Gerontologist. 2011 Apr;51(2):261-72. doi: 10.1093/geront/gnq097. Epub 2011 Jan 17. PMID 21242317
- [Background] Bass DM, Judge KS, Snow AL, Wilson NL, Morgan R, Looman WJ, McCarthy CA, Maslow K, Moye JA, Randazzo R, Garcia-Maldonado M, Elbein R, Odenheimer G, Kunik ME. Caregiver outcomes of partners in dementia care: effect of a care coordination program for veterans with dementia and their family members and friends. J Am Geriatr Soc. 2013 Aug;61(8):1377-86. doi: 10.1111/jgs.12362. Epub 2013 Jul 19. PMID 23869899
- [Background] Bass DM, Judge KS, Snow AL, Wilson NL, Morgan RO, Maslow K, Randazzo R, Moye JA, Odenheimer GL, Archambault E, Elbein R, Pirraglia P, Teasdale TA, McCarthy CA, Looman WJ, Kunik ME. A controlled trial of Partners in Dementia Care: veteran outcomes after six and twelve months. Alzheimers Res Ther. 2014 Feb 28;6(1):9. doi: 10.1186/alzrt242. eCollection 2014. PMID 24764496
- [Background] Bass DM, Clark PA, Looman WJ, McCarthy CA, Eckert S. The Cleveland Alzheimer's managed care demonstration: outcomes after 12 months of implementation. Gerontologist. 2003 Feb;43(1):73-85. doi: 10.1093/geront/43.1.73. PMID 12604748

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Veterans and caregivers were considered enrolled (N = 144 total participants), and are reported here as dyads. Enrollment numbers in this section refers to dyads/ caregivers. (Veteran participants with dementia were not enrolled without a caregiver, but a caregiver could be enrolled without a participating person with dementia.) N = 4 caregivers were enrolled (completed informed consent) but did not complete baseline assessment and therefore were not randomized to group.
Groups:
- Care Consultation (CC): Care Consultation (CC): is an established telephone-based, empowerment intervention that uses coaching and emotional support to mobilize family caregivers and individuals with dementia through psychoeducation, resource referral, psychosocial support, and encouragement of informal and formal service use utilization. A computerized clinical tool called the Care Consultation Information System (CCIS) guides the delivery of protocol components. Rather than a strong focus on assessment, this intervention is designed to quickly identify areas of unmet need through brief trigger questions called the "initial assessment" - much like an interview guide - which then immediately shapes development of concrete action plans.
  Care Consultation (CC): Care Consultation (CC): is an established telephone-based, empowerment intervention that uses coaching and emotional support to mobilize family caregivers and individuals with dementia through psychoeducation, resource referral, psychosocial support, and encouragement of informal and formal service use utilization. A computerized clinical tool called the Care Consultation Information System (CCIS) guides the care consultant through a standardized delivery of protocol components. Rather than a strong focus on assessment, this intervention is designed to quickly identify areas of unmet need through brief trigger questions called the "initial assessment," which then immediately shapes development of concrete action plans.
- Care Consultation + Counseling (CC+C): Care Consultation + Counseling (CC+C): is consistent with the original CC protocol in that the therapist partners with each dyad in a patient-centered way to prioritize unmet needs as identified during the CC initial assessment. Once this phase has been completed, typically within the first 2 sessions, the CC+C therapist will determine when to initiate counseling sessions targeting 8-10 domains of potential distress (grief, hostility, sexual intimacy, etc.). The counseling component of the CC+C intervention incorporates elements of existing manualized interventions that have been tailored for this population and follow a cognitive behavioral therapy framework.
  Counseling (C): The counseling component is tailored for this population and follow a cognitive behavioral therapy framework. Counseling sessions will be completed for 8-10 domains of potential distress (grief, hostility, sexual intimacy, etc.).
Period: Overall Study
Arm/Group | Care Consultation (CC) | Care Consultation + Counseling (CC+C)
Started (Dyads at Baseline in the CC group included n = 40 Caregivers and n = 32 Veterans with dementia. Dyads at Baseline in the CC+C group included n = 42 Caregivers and n = 30 Veterans with dementia.) | 40 | 42
Completed (Dyads at 6-months in the CC group included n = 28 Caregivers and n = 17 Veterans with dementia. Dyads at 6-months in the CC+C group included n = 26 Caregivers and n = 16 Veterans with dementia.) | 28 | 26
Not Completed | 12 | 16
Not completed — Lost to Follow-up | 8 | 8
Not completed — Withdrawal by Subject | 4 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Care Consultation (CC) | Care Consultation + Counseling (CC+C) | Total
Number analyzed (Participants) | 40 | 42 | 82
Age, Continuous [Mean (Full Range); unit: years] | 65.34 [46 to 91] | 64.68 [26 to 86] | 65.00 [26 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 37 | 73
  Male | 4 | 5 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 40 | 42 | 82
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 14 | 27
  White | 26 | 28 | 54
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40 | 42 | 82

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Caregiver Burden Scores on the Zarit Caregiver Burden Inventory
Description: The Zarit Caregiver Burden Inventory is a measure of strain related to providing care for someone with dementia. Scores range from 0 to 48 with higher scores indicating more caregiver burden.
Time Frame: Baseline, 6 months
Population: Statistics control for covariates that were different between the two groups at baseline (i.e., Montreal Cognitive Assessment, MoCA, and education); analyses are based on all cases with valid data for all variables in the model. Number of participants in this section refers to caregivers.
Measure: Mean (Standard Deviation); unit: change units on a scale
Arm/Group | Care Consultation (CC) | Care Consultation + Counseling (CC+C)
Number analyzed (Participants) | 21 | 18
change units on a scale | -2.38 (6.77) | 0.22 (5.26)
Statistical Analysis 1: Comparison: Care Consultation (CC) vs Care Consultation + Counseling (CC+C); Test type: Superiority; p = .483, ANCOVA; Caregiver education, cognitive status of the person with dementia, and baseline caregiver burden scores were included in the model as covariates

2. Primary Outcome: Change From Baseline in Relationship Cohesion on the Dyadic Adjustment Scale
Description: Relationship satisfaction and cohesion measure for spouses and partners in a romantic relationship. Scores range from 0 to 151, and higher scores indicate higher levels of relationship satisfaction. Not all caregivers were in a romantic relationship with the person with dementia, this scale was only administered to dyads who were married or partnered (e.g., adult children caregivers would not have received this measure).
Time Frame: Baseline, 6 months
Population: Number of participants refers to number of spousal caregivers/ caregivers in a romantic relationship with the Veteran/ person with dementia.
Measure: Mean (Standard Deviation); unit: change units on a scale
Arm/Group | Care Consultation (CC) | Care Consultation + Counseling (CC+C)
Number analyzed (Participants) | 9 | 11
change units on a scale | 6.44 (21.45) | -2.64 (18.72)
Statistical Analysis 1: Comparison: Care Consultation (CC) vs Care Consultation + Counseling (CC+C); Only caregivers that were currently or previously in a romantic relationship (e.g., spouses, partners) with the person with dementia reported on the Dyadic Adjustment Scale (i.e., N = 20, n = 9 in CC group and n = 11 in CC+C group); Test type: Superiority; p = 0.169, ANCOVA; Caregiver education, cognitive status of the person with dementia, and baseline Dyadic Adjustment Scale scores were included as covariates

3. Primary Outcome: Change From Baseline in Quality of Life on the World Health Organization (WHO) Quality of Life Measure
Description: Change in shared pleasant events, social engagement, and quality of life is hypothesized to be greater in caregivers assigned to CC+C than in CC alone at 6 months. Scores range from 19 to 95, and higher scores indicate better quality of life.
Time Frame: Baseline, 6 months
Population: Statistics control for covariates that were different between the two groups at baseline (i.e., Montreal Cognitive Assessment, MoCA, and education); analyses are based on all cases with valid data for all variables in the model. Number of participants for this outcome measure refers to number of caregivers.
Measure: Mean (Standard Deviation); unit: change units on a scale
Arm/Group | Care Consultation (CC) | Care Consultation + Counseling (CC+C)
Number analyzed (Participants) | 17 | 15
change units on a scale | .59 (5.34) | -2.97 (3.74)
Statistical Analysis 1: Comparison: Care Consultation (CC) vs Care Consultation + Counseling (CC+C); Test type: Superiority; p = 0.763, ANCOVA; Baseline quality of life scores, education, and cognitive status were included as covariates in the model

4. Primary Outcome: Change From Baseline Depressive Symptoms on the Cornell Scale for Depression in Dementia
Description: Depression symptoms measure, scores range from 0 to 38 with higher scores indicating more depressive symptoms as rated by their caregiver.
Time Frame: Baseline, 6 months
Population: Statistics control for covariates that were different between the two groups at baseline (i.e., Montreal Cognitive Assessment, MoCA, and education); analyses are based on all cases with valid data for all variables in the model. Number of participants in this outcome measure refers to number of Veterans with dementia who had scores reported on CSDD at both time points.
Measure: Mean (Standard Deviation); unit: change in units on a scale
Arm/Group | Care Consultation (CC) | Care Consultation + Counseling (CC+C)
Number analyzed (Participants) | 9 | 10
change in units on a scale | -2.000 (5.172) | -1.100 (6.740)
Statistical Analysis 1: Comparison: Care Consultation (CC) vs Care Consultation + Counseling (CC+C); Test type: Superiority; p = 0.780, ANCOVA; Baseline depression scores, cognitive status scores (i.e., MoCA), and education were included in the model as covariates

5. Secondary Outcome: Number and Percentage of Veterans With Dementia in Long-term Care Facilities as Reported by the Caregivers at 12 Months
Description: Number and percentage of Veterans with dementia in long-term care facilities as reported by the caregivers at 12 months.
Time Frame: 12 months
Population: Number of participants in this outcome measure refers to the number of Veterans with dementia in long term care (as reported by the caregivers).
Measure: Count of Participants; unit: Participants
Arm/Group | Care Consultation (CC) | Care Consultation + Counseling (CC+C)
Number analyzed (Participants) | 28 | 26
Participants | 3 | 3

ADVERSE EVENTS:
Time Frame: 1 year
Description: Adverse events include: hospitalizations, emergency room visits, and one participant who had a house fire during the 12-month study period. Reporting of adverse events is based on all caregivers (n = 82) and veterans (n = 62) that were enrolled and randomized; the caregivers and veterans in each group were n = 72 for CC and n = 72 for CC+C, for a total of N = 144 participants.
Arm/Group | Care Consultation (CC) | Care Consultation + Counseling (CC+C)
All-Cause Mortality (participants affected / at risk) | 3/72 | 0/72
Serious Adverse Events (participants affected / at risk) | 11/72 | 10/72
Other Adverse Events (participants affected / at risk) | 1/72 | 0/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Care Consultation (CC) (N=72) | Care Consultation + Counseling (CC+C) (N=72)
Hospitalizations and Emergency Room Visits (Surgical and medical procedures) | 10 (10) | 10 (10)
House fire (Social circumstances) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Care Consultation (CC) (N=72) | Care Consultation + Counseling (CC+C) (N=72)
Duplicate measures collected (Social circumstances) | 1 (1) | 0 (0) — The research team inadvertently collected 12-month assessment measures more than once for one participant.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-13): https://cdn.clinicaltrials.gov/large-docs/32/NCT02585232/Prot_SAP_000.pdf